CLINICAL TRIAL: NCT06319742
Title: Extracellular Vesicle Surface Markers In Acute Cerebrovascular Syndromes.
Acronym: ElViS-ACS
Status: Recruiting | Type: Observational
Sponsor: Ospedale Civico, Lugano (Other Government)
Responsible Party: Principal Investigator, Dr. med. Carlo Cereda, Prof. Dr. med., Ospedale Civico, Lugano
Other Study IDs: NSISTRCR_2201
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Stroke, TIA, Stroke-mimics, Stroke Biomarkers
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stroke
  Interventions: Diagnostic Test: Extracellular vescicles (EV) analysis
- TIA
  Interventions: Diagnostic Test: Extracellular vescicles (EV) analysis
- Stroke Mimic
  Interventions: Diagnostic Test: Extracellular vescicles (EV) analysis

INTERVENTIONS:
Diagnostic Test: Extracellular vescicles (EV) analysis — The patients undergo a blood sample for EV analyses: EVs will be characterized by nanoparticle tracking analysis, western blot, bead-based flow cytometry (direct and inverse approach), and ELISA.
  We will evaluate diameter and concentration of serum nanoparticles (NPs) by nanoparticle tracking analysis (NTA) using NanoSight LM10. Western Blot analysis will be performed on protein lysate after EV immuno-capture (using beads covered with antibodies against EV specific tetraspanins, CD9, CD63 and CD81). EV profiling will be performed using a standardized multiplex bead-based flow cytometric assay, using MACSPlex Human Exosome Kit (Miltenyi Biotec; Bergisch Gladbach, Germany), as previously described. 22 The detection of 37 different surface antigens commonly expressed on EV membrane (including markers from activated platelets, endothelium, and inflammatory cells) will be simultaneously performed.

SUMMARY:
Clinical implication of eventual blood biomarkers for stroke diagnosis and prognosis would be limited, mainly because clinical evaluation and scales (providing stroke severity) or neuroimaging (providing accurate size of the lesion) are more reliable predictors for clinical outcome prediction. In clinical practice, it would be more useful to find a biomarker, which can help to orientate the physician in conditions in which the clinical picture and imaging provide a limited support.

Transient Ischemic Attacks (TIAs) represent a classical example for which a biomarker would be of interest to confirm and distinguish a brain ischemic process from a stroke mimic. Diagnostic biomarkers of TIA have been investigated, but none of the potential candidates reached enough accuracy for TIA diagnosis. Our group has found that Extracellular Vesicles (EVs) could be useful as biomarkers for detecting brain ischemia in patients with TIA because the EV-surface antigen profile appears to be different in patients with transient symptoms, adjudicated to be very likely caused by brain ischemia, compared to patients whose symptoms were less likely to due to brain ischemia. Our study has raised interest in the scientific community recognizing the promising role of of blood-derived EVs analysis in expanding the possibilities to correctly diagnose and classify TIA and stroke events, discriminate them from TIA or stroke mimics, with important future implications in management and therapy of the patients with acute ischemic cerebrovascular syndrome. the validity of our approach needs to be tested in a larger, prospective, multicenter study.

DETAILED DESCRIPTION:
Characterization of extracellular vesicles Extracellular vesicles (EVs) will be characterized in pre-cleared serum samples (see transfer and managements of blood samples). EVs will be characterized by nanoparticle tracking analysis, western blot, bead-based flow cytometry (direct and inverse approach), and ELISA.

We will evaluate diameter and concentration of serum nanoparticles (NPs) by nanoparticle tracking analysis (NTA) using NanoSight LM10 (Malvern Instruments, United Kingdom) equipped with a 405 nm laser and Nanoparticle Tracking Analysis NTA 2.3 analytic software. A camera will record Brownian movement of EVs and size and number of EVs per mL will be calculated by Stokes-Einstein equation. Three videos of 60 s will be recorded for each analysis.

Western Blot analysis will be performed on protein lysate after EV immuno-capture (using beads covered with antibodies against EV specific tetraspanins, CD9, CD63 and CD81). Blots of representative samples will be incubated with primary antibodies against specific markers expressed on the surface or within EVs (TSG101, Syntenin-1, CD81, Alix) and potential contaminants (GRP94, Apolipoprotein A1, Apolipoprotein B48).

EV profiling will be performed using a standardized multiplex bead-based flow cytometric assay, using MACSPlex Human Exosome Kit (Miltenyi Biotec; Bergisch Gladbach, Germany), as previously described. 22 The detection of 37 different surface antigens commonly expressed on EV membrane (including markers from activated platelets, endothelium, and inflammatory cells) will be simultaneously performed. Background will be subtracted from the MFI value of each marker, and then normalized using by the mean fluorescence intensity levels (MFI) of CD9, CD63, and CD81. Levels of expression will be reported as normalized MFI (nMFI; %) for each EV-surface antigen (median value and interquartile range).

After an initial screening by multiplexed assay, single candidate EV biomarkers will be confirmed by either reverse flow cytometry and ELISA techniques.

The reverse flow cytometric assay will be performed by isolating EVs by capture beads coated with antibodies against CD9-CD63-CD81 (EpCam; JSR Micro) and then incubated with fluorochrome-conjugated antibodies against single EV surface antigens, associated to patient diagnosis during the initial screening by MACSPlex assay. Beads incubated with isotype-matched antibodies, and beads incubated in absence of vesicles will serve as controls. Candidate EV biomarkers will be confirmed also by ELISA technique, using specific antibodies as per manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

Affected by:

I. Suspect ischemic minor stroke (acute loss of focal cerebral function of presumed vascular etiology and NIHSS ≤327, 28) within 48 hours of symptoms onset or II. TIA (defined as the acute onset of focal neurological symptoms lasting <24 h and presumed to be caused by brain ischemia at the time of referral)19 III. Symptoms mimicking I. or II. with but with high suspition of a non-ischemic condition being the cause of the event;

2) age ≥18 years; 3) if cerebral magnetic resonance imaging will be performed within 48-72 hours from admission; 4) if baseline CT/MRI is without hemorrhage; 5) if informed consent obtained.

Exclusion Criteria:

1. ocular TIA (amaurosis fugax);
2. contraindications for MRI;
3. pregnancy;
4. concomitant acute/chronic inflammatory disease (e.g., infections, autoimmune disease);
5. concomitant hematological diseases;
6. Central Nervous System infection within 30 days;
7. serious head trauma within 30 days;
8. major surgery within 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll all patients admitted to the stroke Units because of symptoms suggesting a cerebrovascular syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
TIA differentiation from TIA mimics | 72 hours from symptoms onset
  determine the performance of EV profiling (analysis of antigens expressed on vesicles surface), added to a structured clinical (PREDISC score) and imaging evaluation (brain MRI), to discriminate TIAs from TIA mimics (non ischemic events).

SECONDARY OUTCOMES:
TIA differentiation from Stroke | acute phase, 3 and 12 months
  determine the performance of EV profiling to differentiate between TIAs (with negative MRI for acute lesion) and acute ischemic strokes (AIS, MRI confirmed).
Stroke etiology | acute phase, 3 and 12 months
  determine the performance of EVs profiling to categorize pre-specified causes of ischemic events

CONTACTS AND LOCATIONS:
Locations (1):
- Neurocenter of Southern Switzerland, Ospedale Civico, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No